CLINICAL TRIAL: NCT04307537
Title: POIROT TRIAL: Post-Operative Imaging After Urethroplasty With Peri-catheter Retrograde Urethrography Or Trial of Voiding With Voiding Cysto-urethrography
Brief Title: Post-Operative Imaging After Urethroplasty With Peri-catheter Retrograde Urethrography Or Trial of Voiding With Voiding Cysto-urethrography
Acronym: POIROT
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: B670201942454
Record Dates: First submitted 2020-03-04; First posted 2020-03-13 (Actual); Last update posted 2023-01-04 (Actual); Status verified 2023-01

CONDITIONS: Urethral Stricture
MeSH Terms: conditions — Urethral Stricture

STUDY DESIGN:
Intervention Model Description: Within patient comparison
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- pcRUG (Experimental): Peri-catheter retrograde urethrography
  Interventions: Procedure: Post-urethroplasty urethrography
- VCUG (Active Comparator): Voiding cysto-urethrography
  Interventions: Procedure: Post-urethroplasty urethrography

INTERVENTIONS:
Procedure: Post-urethroplasty urethrography — Imaging of the urethra after reconstructive surgery to identify contrast leakage (no, insignificant, signficant).

SUMMARY:
After a reconstructive procedure of the urethra, a transurethral catheter is usually left in place to allow adequate healing of the tissues without exposure to urine. After 7-21 days, depending on several variables (e.g. type of reconstruction, stricture etiology, …), removal of the transurethral catheter is foreseen. However, in order to do so, the clinician first wants to objectify whether the urethra has indeed healed sufficiently and therefore he/she can rely on early postoperative imaging.

Up until today, there is no clear standard about when and how to do early postoperative imaging and current practices are mainly based on expert opinion and habit. Basically, two strategies can be found amongst different urethroplasty centers: peri-catheter retrograde urethrography (pcRUG) and voiding cysto-urethrography (VCUG). A pcRUG is performed by placing a small caliber tube (e.g. feeding tube 5 Fr) in the meatus urethrae of the patient, next to the transurethral catheter (which remains in place), and injecting contrast alongside the catheter. With a VCUG, contrast is injected through the transurethral catheter, up to the bladder. Thereafter, the catheter is removed and the patient is asked to urinate and thus to pass contrast through the urethra.

The primary end-point of this study is to compare 'the rightful decision to maintain the catheter at the time of imaging' between pcRUG only and pcRUG followed by VCUG in a within-patient fashion.

DETAILED DESCRIPTION:
After a reconstructive procedure of the urethra, a transurethral catheter is usually left in place to allow adequate healing of the tissues without exposure to urine. After 7-21 days, depending on several variables (e.g. type of reconstruction, stricture etiology, …), removal of the transurethral catheter is foreseen. However, in order to do so, the clinician first wants to objectify whether the urethra has indeed healed sufficiently and therefore he/she can rely on early postoperative imaging.

Up until today, there is no clear standard about when and how to do early postoperative imaging and current practices are mainly based on expert opinion and habit. Basically, two strategies can be found amongst different urethroplasty centers: peri-catheter retrograde urethrography (pcRUG) and voiding cysto-urethrography (VCUG). A pcRUG is performed by placing a small caliber tube (e.g. feeding tube 5 Fr) in the meatus urethrae of the patient, next to the transurethral catheter (which remains in place), and injecting contrast alongside the catheter. With a VCUG, contrast is injected through the transurethral catheter, up to the bladder. Thereafter, the catheter is removed and the patient is asked to urinate and thus to pass contrast through the urethra.

In both of the aforementioned imaging modalities, patients are installed similarly on the X-ray table and an antero-posterior X-ray image is made1. In patients with no or insignificant, wisp-like extravasation of contrast, the transurethral catheter can safely be removed. In case of significant contrast extravasation, as defined by Grossgold et al., the catheter is maintained or replaced for another week and one week later, imaging is repeated2.

Both pcRUG and VCUG are not perfect and involve a number of flaws. The main issue with pcRUG is represented by the potential impact of several variables on the image: different levels of pressure in the urethra by different strength of injection, different calibers of tubes through which the contrast is injected, etc. As regards VCUG, an important amount of patients does not achieve to void while being on the X-ray table, which can lead to a long duration of the procedure or even no imaging at all. Another important problem is the fact that if the patient has a significant extravasation of contrast, the catheter needs to be replaced through the freshly reconstructed, and apparently still leaking, urethra. This may be difficult and is often bothersome for the patient.

Given the drawbacks mentioned above, a combination of both techniques can be administered to overcome the flaws of each separate imaging modality and could as such be considered the standard of care in early postoperative imaging after urethroplasty. However, the combination of both techniques includes a higher exposure to radiation than one separate technique and one could wonder what the added value of VCUG after pcRUG is and whether or not this is worth the extra exposure to radiation. To date, there is no such data and a wide variability of strategies is used in the different urethroplasty practices worldwide.

Against this background, the primary end-point of this study is to compare 'the rightful decision to maintain the catheter at the time of imaging' between pcRUG only and pcRUG followed by VCUG in a within-patient fashion.

ELIGIBILITY:
Inclusion Criteria:

* Voluntarily signed written informed consent according to the rules of Good Clinical Practice (Declaration of Helsinki) and national regulations (Appendix B).
* Age ≥ 18 years.
* Male patient.
* Anterior urethral stricture disease (penile, bulbar, penobulbar and panurethral strictures are allowed).
* Procedure was ended with leaving a transurethral catheter in place with foreseen catheter removal and early postoperative imaging after x days.

Exclusion Criteria:

* Absence of signed written informed consent (Appendix B).
* Age < 18 years.
* Female patients.
* Transgender patients.
* Posterior urethral stenosis
* Bladder neck reconstruction
* Patients in which no catheter has been left in place at the end of the procedure.
* Patients in which there is no need for early postoperative imaging, upon discretion of the treating clinician.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2020-01-21 (Actual); Primary Completion 2021-09-01 (Actual); Study Completion 2021-09-01 (Actual)

PRIMARY OUTCOMES:
Percentage of 'rightful decision to maintain the catheter at the time of imaging' between pcRUG only and VCUG. | 1 day (day of original investigation)
  In other words, the amount of catheters maintained during the investigation divided by the number of significant extravasations requiring perpetuated catheter stay.

SECONDARY OUTCOMES:
Difference in radiation exposure between pcRUG and VCUG expressed in mGy/(cm*cm) | 1 day (moment of original investigation)
  Difference in dose of radiation exposure will be assessed with the Mann-Whitney U-test.
Difference in the amount of significant extravasations that is picked up with pcRUG versus VCUG. | Results of both pcRUG and VCUG will be shown to the treating clinician at least 4 weeks after the original investigation and the clinician will have to choose between 'no or insignificant contrast leakage' versus 'significant contrast leakage'.
  Results of both pcRUG and VCUG will be shown to the treating clinician at least 4 weeks after the original investigation and the clinician will have to choose between 'no or insignificant contrast leakage' versus 'significant contrast leakage'.
Intra-observer variability of both pcRUG and VCUG | First blinded assessment (at least 4 weeks after original investigation) versus second blinded assessment another 4 weeks later.
  Reproducibility will be assessed with intraclass correlation coefficients. A threshold of >0.70 will be used as threshold for good intraclass correlation and thus good reproducibility.
Inter-observer variability of both pcRUG and VCUG | Two experienced clinicians will be compared regarding decision making during the first blinded assessment (at least 4 weeks after the original investigation).
  Inter-observer variability will be assessed with Cohen's kappa. A threshold of >0.70 will be used for good inter-observer variability
Amount of patients unable to void while being on the X-ray table | 1 day (moment of original investigation)
  During VCUG, patients have to void after catheter removal to allow urethral imaging. Often, patients are unable to void while on the X-ray table.

CONTACTS AND LOCATIONS:
Locations (1):
- Dept. of Urology, Ghent University Hospital, Ghent, East-Flanders, Belgium

IPD SHARING:
Plan to Share IPD: Undecided